CLINICAL TRIAL: NCT00433784
Title: Evaluation of the Effect of the H2 Haplotype and CYP3As Polymorphisms on the Antiplatelet Response to Clopidogrel Given Before Elective Percutaneous Coronary Intervention
Brief Title: H2 Haplotype and CYP3As Polymorphisms and the Antiplatelet Response to Clopidogrel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: C.E.2004-06-24
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2008-06

CONDITIONS: Coronary Artery Disease; Elective Percutaneous Coronary Intervention
Keywords: clopidogrel; platelet aggregation; CYP3A; H2 haplotype; polymorphisms
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel
Procedure: Blood sampling - platelet aggregation
Procedure: Blood sampling - genotyping

SUMMARY:
The purpose of this study was to assess whether interpatient variability in the platelet response to clopidogrel is partly due to polymorphisms of the hepatic cytochrome P450 (CYP450)3A and of the clopidogrel-P2Y12 receptor genes.

DETAILED DESCRIPTION:
Clopidogrel owes its antiplatelet effect to irreversible inhibition of the purinergic platelet receptor, P2Y12. It is estimated that approximately 4%-30% of patients treated with conventional doses of clopidogrel do not display adequate platelet response. Moreover, patients with low response to clopidogrel may be at higher risk for atherothrombotic events. Clopidogrel, being a prodrug, requires oxidation by the hepatic cytochrome P450 (CYP450)3A to generate an active metabolite.The level of CYP3A4 activity has been shown to correlate with the inhibitory effect of clopidogrel on platelet aggregation in healthy volunteers. However, CYP3As expression and activity vary among individuals. It is estimated that most of this variability is caused by individual genetic makeup.Polymorphisms of the P2Y12 receptor may also play a role in the variability in clopidogrel response. The P2Y12-H2 haplotype was associated with higher maximal platelet aggregation in response to adenosine diphosphate (ADP) as compared to the P2Y12-H1 haplotype probably due to an increase in the number of receptors on the platelet surface. It has also been suggested that carriers of the H2 haplotype might be at higher risk of developing peripheral artery disease.

Comparisons: Presence of CYP3A5 polymorphism and of the H2 haplotype compared to absence of these polymorphisms on the antiplatelet response to clopidogrel across a wide range of clopidogrel dosing regimens in patients with suspected or demonstrated coronary artery disease (CAD) scheduled to undergo elective percutaneous coronary intervention (PCI).

Platelet aggregation was measured by optical aggregometry with (ADP) 20 μmol/L as the agonist in patients before clopidogrel initiation and at the time of diagnostic coronary angiography. Genotyping was performed by standard polymerase chain reaction (PCR) method to identify expressors of CYP3A5 and P2Y12 H2 haplotype carriers.

ELIGIBILITY:
Inclusion Criteria:

* Documented coronary artery disease (CAD) requiring an elective diagnostic coronary angiography with or without percutaneous coronary intervention (PCI)

Exclusion Criteria:

* Major bleeding disorders or active bleeding;
* Acute MI within 14 days of recruitment;
* Unstable angina with ST-segment changes of > or = 1 mm in at least two contiguous electrocardiographic leads at rest, a troponin level of > 0.06 ug/L or both within 14 days of recruitment;
* Stroke within the last 3 months;
* Platelet count < 100 x 109/L;
* Prothrombin time > 1.5 times control;
* Hematocrit < 25% or hemoglobin level < 100 g/L;
* Alcohol or drug abuse;
* Enrolment in other investigational drug trials within the previous month;
* Use of thienopyridines, glycoprotein (GP) IIb/IIIa inhibitors, warfarin or acenocoumarol within the prior week;
* Allergic reaction or any contraindication to clopidogrel or aspirin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-09; Study Completion 2006-04

PRIMARY OUTCOMES:
Effect of CYP3A5 polymorphisms and of the H2 haplotype on the inhibitory effect of clopidogrel on platelet aggregation at the time of diagnostic coronary angiography as measured by optical aggregometry with adenosine diphosphate (ADP) 20 μmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Jean G Diodati, MD, Principal Investigator — Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Locations (1):
- Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec, Canada